CLINICAL TRIAL: NCT05738330
Title: Comparative Effectiveness of Two Approaches to Symptom Monitoring in Hemodialysis
Brief Title: Symptom Monitoring in Hemodialysis
Acronym: SMaRRT-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Duke University (Other); University of New Mexico (Other); Fresenius Medical Care North America (Industry); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Laura Dember, MD, Professor of Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 852661
Record Dates: First submitted 2023-01-31; First posted 2023-02-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: End Stage Kidney Disease
Keywords: End stage kidney disease; Kidney; Hemodialysis; Dialysis; Symptom monitoring; Electronic Patient-Reported Outcome Measure (ePROM)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: The design is a multi-center cluster-randomized trial with randomization performed at the level of the dialysis clinic. Dialysis clinics will be assigned to either the SMaRRT-HD group (18 clinics) or the Usual Care group (18 clinics). SMaRRT-HD is a symptom monitoring system that includes 1) tablet-based symptom reporting using a patient reported outcome measure (PROM) and 2) supported clinician follow-up consisting of symptom alerts, symptom management guidance, and tracking reports to share with patients. Dialysis clinics assigned to Usual Care will not use SMaRRT-HD or any other trial-driven procedures. Usual Care clinics will monitor symptoms through clinical interactions with participants and by administering a HRQOL survey. The trial uses a hybrid Type 1 effectiveness-implementation approach with effectiveness of the intervention assessed with patient-reported outcomes and biomedical outcomes, and implementation assessed with integrated qualitative and quantitative outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMaRRT-HD (Symptom Monitoring on Renal Replacement Therapy - Hemodialysis) (Active Comparator): Dialysis clinics randomized to SMaRRT-HD will implement the SMaRRT-HD symptom monitoring system. SMaRRT-HD consists of 1) tablet-based symptom reporting using a patient reported outcome measure (PROM) and 2) supported clinician follow-up consisting of symptom alerts, guidances for symptom management, and symptom tracking reports that are shared with patients. For trial participants in SMaRRT-HD clinics, the SMaRRT-HD system will be implemented in addition to the Usual Care approach to symptom monitoring.
  Interventions: Behavioral: Symptom Monitoring on Renal Replacement Therapy - Hemodialysis (SMaRRT-HD)
- Usual Care (Active Comparator): Dialysis clinics randomized to Usual Care will not adopt SMaRRT-HD or any other trial-driven procedures. Usual Care clinics will monitor symptoms through clinical care interactions with participants and by administering a CMS-mandated Health-Related Quality of Life (HRQOL) survey that includes questions about symptoms.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Symptom Monitoring on Renal Replacement Therapy - Hemodialysis (SMaRRT-HD) — Dialysis clinics randomized to the SMaRRT-HD group will use the SMaRRT-HD system to capture patient-reported symptoms and support clinician follow-up. The online system includes the patient symptom ePROM surveys, clinician real-time email alerts, clinician guidances for symptom management, and patient-facing symptom reports as well as an administrative dashboard supporting management of trial participants at clinics using SMaRRT-HD. Designated clinic personnel (i.e., patient care technicians and nurses) will receive training on how to use the system to administer the symptom ePROM surveys to patients on tablet computers. Designated clinic nurses and medical providers will receive training on how to access guidances for symptom management and patient-facing symptom reports in the SMaRRT-HD system. For trial participants in SMaRRT-HD clinics, the SMaRRT-HD system will be implemented in addition to the Usual Care approach to symptom monitoring.
  Arms: SMaRRT-HD (Symptom Monitoring on Renal Replacement Therapy - Hemodialysis)
Behavioral: Usual Care — Dialysis clinics randomized to Usual Care will not adopt SMaRRT-HD or any other trial-driven procedures. Usual Care clinics will monitor symptoms through clinical care interactions with participants and by administering a CMS-mandated Health-Related Quality of Life (HRQOL) survey that includes questions about symptoms.
  Arms: Usual Care

SUMMARY:
The SMaRRT-HD trial is a cluster randomized trial of symptom monitoring with supported clinician follow-up using the SMaRRT-HD electronic patient reported outcome measure (ePROM) system versus Usual Care. Approximately 2400 patients at up to 36 geographically and racially diverse US hemodialysis clinics will be enrolled. The primary trial hypothesis is that regular symptom patient reported outcome measure (PROM) administration with supported clinician follow-up in dialysis care will reduce suffering and improve outcomes by prompting treatment of unrecognized symptoms, and enhancing patient-care team communication. Clinics randomized to the SMaRRT-HD group will adopt the use of SMaRRT-HD for 12 months. SMaRRT-HD is a symptom monitoring system that includes 1) tablet-based symptom reporting using a PROM and 2) supported clinician follow-up consisting of symptom alerts, guidances for symptom management, and symptom tracking reports that are shared with patients. Dialysis clinics randomized to Usual Care will not adopt SMaRRT-HD or any other trial-driven procedures. Usual Care clinics will monitor symptoms through clinical care interactions with participants and by administering a Health Related Quality of Life survey that includes questions about symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Treatment with hemodialysis at a participating dialysis clinic
* English or Spanish speaking

Exclusion Criteria:

* Not willing to report their symptoms using the SMaRRT-HD platform
* Not willing to share clinically acquired data with the research team
* Underlying condition such as dementia that is anticipated to prevent comprehension of the trial information document (fact sheet)
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Severity of dialysis-associated symptoms (Effectiveness) | Baseline, 6 months, 12 months
  This outcome will be assessed as change in the Dialysis Symptom Index-Severity Score over 12 months (primary endpoint).
  Participants are asked whether or not they experienced symptoms during the past week. If the response is yes, the participant is asked to indicate "How much did it bother you?". Lowest score - 0; Highest score - 150. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Health-related quality of life (Effectiveness) | Baseline, 6 months, 12 months
  EuroQOL 5D-5L (EQ-5D-5L)
  Participants are asked about 5 different domains that can affect people's quality of life (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression). Participants respond on a scale of 1 to 5 where 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. An EQ-5D summary index is derived by applying a formula (developed by EuroQol Group) that attaches values (weights) to each of the levels in each dimension. A higher score indicates a better outcome.
Post-dialysis recovery time (Effectiveness) | Baseline, 6 months, 12 months
  Recovery time question
Fatigue (Effectiveness) | Baseline, 6 months, 12 months
  PROMIS Fatigue SF 6a
  Fatigue will be measured using the PROMIS Fatigue Short Form (SF) 6a. Normalized score reported as t-values. The full range of possible scores is 26.2 - 65.6. 50 indicates the population mean with a standard deviation of 10. A lower score represents a better outcome.
Pain interference (Effectiveness) | Baseline, 6 months, 12 months
  Brief Pain Inventory (BPI)- Interference
  Participants are asked how much, during the past week, pain has interfered with different activities. This is typically scored as the mean of the seven items. Lowest score - 0; Highest score - 10. A higher score indicates a worse outcome.
Anxiety (Effectiveness) | Baseline, 6 months, 12 months
  Generalized Anxiety Disorder (GAD)-7
  Participants are asked to report how often during the past 2 weeks they have had symptoms or experiences. Lowest score - 0; Highest score - 21. Higher score indicates a worse outcome.
Depression (Effectiveness) | Baseline, 6 months, 12 months
  Patient Health Questionnaire (PHQ)-8
  Participants are asked to report how much during the last 2 weeks they have experienced problems. Lowest score - 0; Highest score - 24. Higher score indicates a worse outcome.
Healthcare Engagement (Effectiveness) | Baseline, 6 months, 12 months
  Healthcare Engagement - Short Form 8a (PHE-8a)
  Participants are asked to respond to statements with how true each statement is for them at the time the questionnaire is administered. Responses range from "Not at all true" to "Very true". The PHE-8a uses item response theory-based scoring converted to standardized T-scores. A higher score indicates a better outcome.
Hospitalizations (Effectiveness) | Duration of active 12 month study participation plus 6 months; 18 months total
  Hospitalization rate
Mortality (Effectiveness) | Duration of active 12 month study participation plus 6 months; 18 months total
  Mortality rate
Missed dialysis sessions (Effectiveness) | Duration of active 12 month study participation
  The number of missed dialysis sessions during participation in the the trial.
Shortened dialysis sessions (Effectiveness) | Duration of active 12 month study participation
  The number of shortened dialysis sessions during participation in the the trial.
Penetration (Implementation) | Duration of active 12 month study participation
  SMaRRT-HD completion rates collected from the SMaRRT-HD system and KDQOL™-36 completion rates collected from the dialysis medical record
Fidelity (Implementation); Clinical action after PROM use; All Clinics | Duration of active 12 month study participation
  Evidence in the dialysis medical record of clinician action in response to a reported symptom.
Fidelity (Implementation); Patient-reported clinician follow-up; All Clinics | Baseline, 6 months, and 12 months
  Patient response to a Computer-Assisted Telephone Interview-administered question about the occurrence of clinician follow-up of a reported symptom.
Fidelity (Implementation); Patient/clinician-reported follow-up activities; All Clinics | 6 months, and 12 months
  Patient, clinic personnel, and medical provider responses to survey questions about the occurrence of clinician follow-up of a reported symptom.
Fidelity (Implementation); Clinician access of symptom guidances; SMaRRT-HD Clinics | Duration of active 12 month study participation
  In SMaRRT-HD clinics only, evidence in the SMaRRT-HD system of clinician access of symptom guidances within 7 days of each administration of the SMaRRT-HD symptom ePROM.
Fidelity (Implementation); Clinician access of symptom reports; SMaRRT-HD Clinics | Duration of active 12 month study participation
  In SMaRRT-HD clinics only, evidence in the SMaRRT-HD system of clinician access of symptom reports within 7 days of each administration of the SMaRRT-HD symptom ePROM.
Fidelity (Implementation); Patient-reported receipt of symptom summary; All Clinics | Baseline, 6 months, and 12 months
  Patient response to a Computer-Assisted Telephone Interview-administered question about the receipt of symptom summaries.
Acceptability (Implementation); Surveys; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to survey questions about the acceptability of patient-dialysis care team communication about symptoms.
Acceptability (Implementation); Interviews; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to interview questions about the acceptability of patient-dialysis care team communication about symptoms.
Acceptability (Implementation); Surveys; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to survey questions about the acceptability of the SMaRRT-HD system components.
Acceptability (Implementation); Interviews; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to interview questions about the acceptability of the SMaRRT-HD system components.
Appropriateness (Implementation); Surveys; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to survey questions about the appropriateness of patient-dialysis care team communication about symptoms.
Appropriateness (Implementation); Interviews; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to interview questions about the appropriateness of patient-dialysis care team communication about symptoms.
Appropriateness (Implementation); Surveys; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to survey questions about the appropriateness of the SMaRRT-HD system components.
Appropriateness (Implementation); Interviews; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to interview questions about the appropriateness of the SMaRRT-HD system components.
Feasibility (Implementation); Surveys; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to survey questions about feasibility of patient-dialysis care team communication about symptoms.
Feasibility (Implementation); Interviews; All Clinics | 6 months and 12 months
  Patient, clinic personnel, and medical provider responses to interview questions about feasibility of patient-dialysis care team communication about symptoms.
Feasibility (Implementation); Interviews; Dialysis provider organization corporate leaders | Interviews will be conducted before the optimization phase and after the end of the trial.
  Corporate leader responses to interview questions about the importance, feasibility, and potential for sustainability of regularly administering PROMs in routine dialysis care.
Feasibility (Implementation); Surveys; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to survey questions about the feasibility of the SMaRRT-HD system components.
Feasibility (Implementation); Interviews; SMaRRT-HD Clinics | 6 months and 12 months
  In SMaRRT-HD clinics only, patient, clinic personnel, and medical provider responses to interview questions about the feasibility of the SMaRRT-HD system components.

OTHER OUTCOMES:
Quality of patient-clinician communication (Effectiveness) | Baseline, 6 months, 12 months
  In-Center Hemodialysis Consumer Assessment of Healthcare Providers and Systems (ICH CAHPS)- Communication and Caring Domain

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Flythe, MD, Principal Investigator — University of North Carolina, Chapel Hill; Laura Dember, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Fresenius Medical Care, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The primary method by which data will be shared with the scientific community will be through peer-reviewed publications and presentations at scientific and professional society meetings. A final report of the research results will be submitted to PCORI for peer review in accordance with the PCORI Peer Review and Findings Release Process. Plain language summaries of the results will be provided to all participating dialysis clinics for distribution to all patients, personnel, and medical providers. Data Sharing will be consistent with PCORI's Policy for Data Management and Data Sharing and as permitted by the project contracts and data use agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Flythe JE, Picataggio CB, Bernardo L, Dalrymple LS, Kossmann RJ, DeWalt DA, Hanson LC, Wang V, Unruh ML, Hsu JY, Dember LM. Design and rationale of the SMaRRT-HD study: A pragmatic, randomized trial of symptom monitoring for individuals receiving maintenance hemodialysis. Contemp Clin Trials. 2025 Oct;157:108058. doi: 10.1016/j.cct.2025.108058. Epub 2025 Aug 30. PMID 40889553